CLINICAL TRIAL: NCT01088594
Title: A Methodological Study To Evaluate The Effects of Single Oral Doses Of Pioglitazone 45 mg And Rosiglitazone 8 mg On Sodium Balance In Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: S337.1.004; 2009-017263-42
Record Dates: First submitted 2010-02-26; First posted 2010-03-17 (Estimated); Last update posted 2010-03-17 (Estimated); Status verified 2010-03

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: urinary sodium excretion; Pioglitazone; Rosiglitazone; Methodological study
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Pioglitazone; Rosiglitazone

ARMS (3):
- 1 (Experimental): pioglitazone 45 mg
  Interventions: Drug: pioglitazone/rosiglitazone/placebo; Drug: rosiglitazone/pioglitazone/placebo; Drug: placebo/pioglitazone/rosiglitazone; Drug: pioglitazone/placebo/rosiglitazone; Drug: rosiglitazone/placebo/pioglitazone; Drug: placebo/rosiglitazone/pioglitazone
- 2 (Experimental): Rosiglitazone 8 mg
  Interventions: Drug: pioglitazone/rosiglitazone/placebo; Drug: rosiglitazone/pioglitazone/placebo; Drug: placebo/pioglitazone/rosiglitazone; Drug: pioglitazone/placebo/rosiglitazone; Drug: rosiglitazone/placebo/pioglitazone; Drug: placebo/rosiglitazone/pioglitazone
- 3 (Placebo Comparator): Placebo
  Interventions: Drug: pioglitazone/rosiglitazone/placebo; Drug: rosiglitazone/pioglitazone/placebo; Drug: placebo/pioglitazone/rosiglitazone; Drug: pioglitazone/placebo/rosiglitazone; Drug: rosiglitazone/placebo/pioglitazone; Drug: placebo/rosiglitazone/pioglitazone

INTERVENTIONS:
Drug: pioglitazone/rosiglitazone/placebo — single oral dose of pioglitazone 45mg + single oral dose of rosiglitazone 8mg +single oral dose of placebo
Drug: rosiglitazone/pioglitazone/placebo — single oral dose of rosiglitazone 8mg + single oral dose of pioglitazone 45mg + single oral dose of placebo
Drug: placebo/pioglitazone/rosiglitazone — single oral dose of placebo + single oral dose of pioglitazone 45mg + single oral dose of rosiglitazone 8mg
Drug: pioglitazone/placebo/rosiglitazone — single oral dose of pioglitazone 45mg +single oral dose of placebo + single oral dose of rosiglitazone 8mg
Drug: rosiglitazone/placebo/pioglitazone — single oral dose of rosiglitazone 8mg + single oral dose of placebo + single oral dose of pioglitazone 45mg
Drug: placebo/rosiglitazone/pioglitazone — single oral dose of placebo + single oral dose of rosiglitazone 8mg + single oral dose of pioglitazone 45mg

SUMMARY:
A single centre, open, randomized, placebo controlled, 3 period cross-over study to evaluate the effects of single oral doses of pioglitazone 45mg, rosiglitazone 8mg and placebo on urinary sodium excretion in 12 healthy male volunteers

ELIGIBILITY:
Inclusion Criteria Volunteers with Body Mass Index 18.0-28.0 kg/m2 Exclusion Criteria Clinically relevant medical history

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2010-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
Time-course urinary sodium excretion calculated on the Day 1 of each study period | 0-6 hours
Time-course absolute urinary sodium excretion calculated on the Day 1 of each study period | 0-6 hours

SECONDARY OUTCOMES:
Sodium clearance on Day 1 of each study period | 0-6 hours
Creatinine clearance calculated on Day 1 of each study period | 0-6 hours

CONTACTS AND LOCATIONS:
Overall Officials: Claire Nee, Study Director — Solvay Pharmaceuticals
Locations (1):
- S337.1.004 Site #, London, United Kingdom